CLINICAL TRIAL: NCT02490085
Title: An Open-label, Randomized, Two-way, Cross-over Multicenter Study to Assess the Efficacy of Closed-loop Strategy as Compared to Multiple Daily Injections in Regulating Glucose Levels During 24 Hours in Adults With Type 2 Diabetes Under Intensive Insulin Therapy
Brief Title: Closed-loop Control of Glucose Levels (Artificial Pancreas) for 24 Hours in Adults With Type 2 Diabetes Under Intensive Insulin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Réseau de recherche en santé cardiométabolique, diabète et obésité (Unknown)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-12
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Closed-loop strategy; Artificial pancreas; Insulin; Elderly; Multiple daily injections; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Hypoglycemia | interventions — Methods; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple daily injections (Active Comparator): Subjects will use multiple daily injections to regulate glucose levels. Subject's usual insulin analog will be used.
  Interventions: Other: 24-hour intervention with multiple daily injections; Drug: Insulin; Device: Dexcom G4 Platinum
- Closed-loop strategy (Active Comparator): Variable subcutaneous insulin infusion rates will be used to regulate glucose levels. Subject's usual fast-acting insulin analog will be infused using a subcutaneous infusion pumps (Accu-Chek Combo, Roche). The glucose level as measured by the real time sensor (Dexcom G4 Platinum, Dexcom) will be entered manually into the computer every 10 minutes. The pumps' infusion rate will then be changed manually based on the computer generated recommendation infusion rates.
  Interventions: Other: 24-hour intervention with closed-loop strategy; Drug: Insulin; Device: Insulin pump Accu-Chek Combo; Device: Dexcom G4 Platinum

INTERVENTIONS:
Other: 24-hour intervention with multiple daily injections — Subjects will be admitted at the research clinical facility at 20:00. A cannula will be inserted into an arm or a hand vein for blood sampling purposes. The subjects will carry on with their normal insulin therapy. Two periods of walking of 15 minutes will be performed at 10:00 and 15:00. Meals will be served at 8:00, 12:00 and 17:00. The CHO content of meals will be adapted to subject's usual CHO intake. Venous blood samples (4 ml each) will be obtained for the measurement of the plasma glucose and insulin. Plasma glucagon and C-peptide will be measured every hour. Blood samples will be drawn every 20 minutes.
  Arms: Multiple daily injections
Other: 24-hour intervention with closed-loop strategy — Subjects will be admitted at the research clinical facility at 20:00. A cannula will be inserted into an arm or a hand vein for blood sampling purposes. A cartridge containing subject's usual fast acting insulin analog will be placed in the insulin pump. Closed-loop strategy will start at 21:00 until 21:00 the next day. Neither basal nor prandial insulin injections will be given. Two periods of walking of 15 minutes will be performed at 10:00 and 15:00. Meals will be served at 8:00, 12:00 and 17:00. The CHO content of meals will be adapted to subject's usual CHO intake. Venous blood samples (4 ml each) will be obtained for the measurement of the plasma glucose and insulin. Plasma glucagon and C-peptide will be measured every hour. Blood samples will be drawn every 20 minutes.
  Arms: Closed-loop strategy
Drug: Insulin — Subject's usual insulin analog will be used.
Device: Insulin pump Accu-Chek Combo — During closed-loop intervention, the Accu-Chek Combo (Roche) insulin pump will be used
  Arms: Closed-loop strategy
Device: Dexcom G4 Platinum — In both visits, glucose levels will be measure with the Dexcom G4 Platinum (Dexcom)

SUMMARY:
The introduction of insulin pump therapy in patients with type 2 diabetes using multiple daily injections and poorly controlled can be considered in order to improve glycemic control. Recent developments of continuous glucose sensors and insulin infusion pumps have motivated the research toward "closed-loop'' strategies to regulate glucose levels for patients with diabetes. In a closed-loop strategy, the pump(s) infusion rate is altered based on a computer generated recommendation that rely on continuous glucose sensor readings. This study confirmed the feasibility and potential of the closed-loop strategy to improve glycemic control while reducing the risk of hypoglycemia in patients with type 2 diabetes but did not target the population most likely to benefit from this strategy.The objective ot this study is to compare the efficacy of closed-loop strategy to multiple daily injections in regulating glucose levels for 24 hours in elderly adults with type 2 diabetes under intensive insulin therapy. The investigators hypothesize that closed-loop strategy will increase the time spent in the target range in adults with type 2 diabetes compared to multiple daily injections.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes.
2. Males and females ≥ 55 years of old.
3. Body mass index above 25 kg/m2
4. Non fragile defined based on Moorhouse et al. scale [23].
5. Using at least 3 insulin injections per day. However, basal insulin injection must be injected at bedtime without injection of basal insulin in the morning. Combination with any other anti-diabetic therapy is acceptable as long at this therapy was introduced at least 6 weeks prior the 1s intervention and is kept stable all along the protocol.
6. HbA1c above 6%.

Exclusion Criteria:

1. Advanced

   1. Nephropathy defined by creatinine clearance <30 ml/min.
   2. Retinopathy as proliferative retinopathy or recent (<3 month) eye bleeding or laser therapy. If the patient have undergone panphoto-coagulation inclusion is acceptable.
   3. Autonomic neuropathy with clinically significant gastroparesis according to investigator evaluation.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. A recent (< 2 months) injury to body or limb, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the ability to walk.
4. A recent (< 2 months) infection needing IV antibiotic or hospitalization
5. Severe hypoglycemic episode within two weeks of screening.
6. Current use of glucocorticoid medication (by any route of administration except low dose stable inhaled).
7. Recent initiation or dose modification (<2 months) of therapy known to interfere with glucose metabolism (e.g. neuroleptics, anti-psychotics, etc.)
8. Known or suspected allergy to the trial products or meal contents.
9. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose concentrations spent in the target range | 24 hours
  The target range is defined as between 4.0 and 10.0 mmol/L 2-hour postprandial and between 4.0 to 8.0 mmol/L otherwise.

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent between 4.0 to 10.0 mmol/L | 24 hours
Percentage of time of plasma glucose levels spent below 4.0 mmol/L | 24 hours
Percentage of time of plasma glucose levels spent below 3.5 mmol/L | 24 hours
Percentage of time of plasma glucose levels spent above 8.0 mmol/L | 24 hours
Percentage of time of plasma glucose levels spent above 10.0 mmol/L | 24 hours
Percentage of time of overnight plasma glucose levels spent below 4.0 mmol/L | 8 hours
Percentage of time of overnight plasma glucose levels spent between 4.0 and 8.0 mmol/L | 8 hours
Percentage of time of overnight plasma glucose levels spent between 4.0 and 10.0 mmol/L | 8 hours
Percentage of time of overnight plasma glucose levels spent below 3.5 mmol/L | 8 hours
Percentage of time of overnight plasma glucose levels above 8.0 mmol/L | 8 hours
Percentage of time of overnight plasma glucose levels above 10.0 mmol/L | 8 hours
Area under the curve of plasma glucose levels below 4.0 mmol/L | 24 hours
Area under the curve of plasma glucose levels below 3.5 mmol/L | 24 hours
Area under the curve of plasma glucose levels above 8.0 mmol/L | 24 hours
Area under the curve of plasma glucose levels above 10.0 mmol/L | 24 hours
Area under the curve of overnight plasma glucose levels below 4.0 mmol/L | 8 hours
Area under the curve of overnight plasma glucose levels below 3.5 mmol/L | 8 hours
Area under the curve of overnight plasma glucose levels above 8.0 mmol/L | 8 hours
Area under the curve of overnight plasma glucose levels above 10.0 mmol/L | 8 hours
Mean glucose levels | 24 hours
Total insulin delivery | 24 hours
Standard deviation of plasma glucose concentrations | 24 hours
Coefficient of variance of plasma glucose concentrations | 24 hours
Number of patients experiencing at least one hypoglycemic event requiring treatment | 24 hours
Number of patients experiencing at least one hypoglycemic event requiring treatment | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec